CLINICAL TRIAL: NCT00288223
Title: Multicenter Non Comparative Phase IV Study on the Safety and Efficacy of Telithromycin 800 mg Per Day for 5 Days in the Treatment of Acute Exacerbation of Chronic Bronchitis in Adults
Brief Title: Telithromycin in Acute Exacerbation of Chronic Bronchitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4022
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Bronchitis, Chronic
MeSH Terms: conditions — Bronchitis, Chronic | interventions — telithromycin

ARMS (1):
- 1 (Experimental): telithromycin
  Interventions: Drug: Telithromycin

INTERVENTIONS:
Drug: Telithromycin — one daily intake of 800 mg (i.e. 2 x 400 mg tablets) per os in a single intake with a meal for 5 days.

SUMMARY:
Study objectives:

* to document the clinical efficacy of telithromycin(800 mg per day for 5 days) at Test Of the Cure (TOC)visit (D12-D19), in acute exacerbation of chronic bronchitis.
* to assess the long-term clinical efficacy of telithromycin by telephone at D25-D35 (V3)
* to assess the safety of telithromycin

ELIGIBILITY:
Inclusion Criteria:

* Outpatients,
* With a documented history of chronic bronchitis defined by one expectoration daily for at least three consecutive months over at least two consecutive years
* Presenting with an evident acute exacerbation of their disease defined by the presence of at least two of Anthonisen's criteria:

  * exacerbation of dyspnea,
  * increase in the expectoration volume,
  * increase in the expectoration purulence,

Exclusion Criteria:

* Acute bronchitis,
* Chronic obstructive pulmonary disease, those having FEV1 value <35% (FEV1: Forced Expiratory Volume in 1 second)
* Suspected pneumonia or bronchial pneumonia,
* Paroxysmal asthma or continuous dyspnea in asthma,
* Cystic fibrosis,
* Active tuberculosis,
* Lung cancer or lung metastasis,
* Severe bronchiectasia,
* Acute respiratory decompensation,
* Chronic respiratory insufficiency associated with resting hypoxemia,
* Patients requiring hospitalization for parenteral antibiotic treatment
* Patients with suspected or known bacterial infection other than study diseases, as well as associated systemic or intra-tracheal antibiotic treatment other than study treatment,
* Participating in another clinical study with any product within 30 days before the inclusion of study
* Known immunosuppression (AIDS and/or CD4+ lymphocytes < 200/mm3, neutropenia <1500/mm3, blood diseases or terminal stage cancer)
* Cardiovasculary, neurologic or other severe diseases interfering with the compliance with study protocol or confusing with results.

Conditions associated with study medications:

* Hypersensitivity against telithromycin , macrolides or any of the excipients,
* Congenital long QT syndrome or family history of congenital long QT syndrome (this possibility should be excluded with normal ECG) or known acquired QT interval prolongation,
* Treatment with CYP3A4 inducers (rifampicin, carbamazepine, phenytoin, phenobarbital, St-John's-wort) within 2 weeks prior to the study inclusion
* Possibility of treatment with ergot alkaloid derivatives, terfenadine, astemizole, pimozide, cisapride, simvastatin, athorvastatin or lovastatin during studies
* Congenital galactosemia, lactase deficiency glucose or galactose malabsorption syndrome,
* Pregnant or lactating women,
* Women with childbearing potential (e.g. ovulating, pre-menopausal or not surgically sterilized) and do not employ any effective contraception method The patients may not participate to the study more than once. The patients who were treated with study drugs previously may not participate to the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percentage of clinical success (cure + improvement) at TOC visit (D12-19),clinical success at TOC visit in at risk sub-populations, clinical success at follow up visit (D25-35), reinfection rates,discontinuation of treatment rates, compliance | D12-D19 (efficacy assessment) and D25-D35 (telephone follow-up)

SECONDARY OUTCOMES:
Safety assessment of telithromycin (Safety will be assessed on the basis of serious and non serious adverse events) | At V3

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)